CLINICAL TRIAL: NCT06386003
Title: Psilocybin-Assisted Massed Cognitive Processing Therapy for Chronic Posttraumatic Stress Disorder: An Open-label Trial
Brief Title: Psilocybin-Assisted Cognitive Processing Therapy for Chronic PTSD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Toronto Metropolitan University (Other); University of Ottawa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-230
Record Dates: First submitted 2024-04-18; First posted 2024-04-26 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Post Traumatic Stress Disorder; PTSD; Chronic PTSD
Keywords: Post Traumatic Stress Disorder; Psilocybin; Cognitive Processing Therapy
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Psilocybin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Single dose of psilocybin 25mg + Massed cognitive processing therapy
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — Participants will receive a single dose of psilocybin 25mg combined with 12 sessions of massed CPT, and 2 psychotherapy sessions related to psilocybin over 7 days.

SUMMARY:
This is an open-label trial evaluating feasibility, tolerability, safety and efficacy of psilocybin assisted cognitive processing therapy for chronic Posttraumatic Stress Disorder (PTSD).

DETAILED DESCRIPTION:
Current front-line treatments for Posttraumatic stress disorder (PTSD) are ineffective for up to half of patients, with serious medical and societal consequences. It is imperative to improve the efficacy of front-line treatment options, such as cognitive processing therapy (CPT). CPT is an effective treatment for PTSD, including when delivered intensively (i.e., multiple sessions over 7 days). However, a substantial proportion of patients continue to meet criteria for PTSD or have residual PTSD symptoms post-treatment. Psilocybin-assisted CPT may be a potential solution, as preliminary evidence supports the potential of psilocybin to alleviate symptoms of PTSD.

Fifteen participants will receive a single dose of psilocybin 25mg combined with 12 sessions of massed CPT, and 2 psychotherapy sessions related to psilocybin over 7 days. Participants will complete clinician-administered scales, self-reported mental health questionnaires, and use a wearable device. After the 1-week interventional period, participants will enter a 12-weeks follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Meet Diagnostic and Statistical Manual-5th edition (DSM-5) criteria for current PTSD with a duration of 6 months or longer assessed by study psychiatrist;
2. Have a Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) score of 50 or higher, indicating moderate to severe PTSD symptoms;
3. Are willing to refrain from taking any psychiatric medications during the study period.

Exclusion Criteria:

1. Are pregnant or nursing, or are women of child bearing potential who are not practicing an effective means of birth control;
2. Have a history of or a current primary diagnosis of psychotic disorder, schizophrenia, delusional disorder, borderline personality disorder, schizoaffective disorder, bipolar disorder or, dissociative identity disorder;
3. Have evidence or history of coronary artery disease or cerebral or peripheral vascular disease, hepatic disease with abnormal liver enzymes, or any other medical disorder judged by the investigator to significantly increase the risk of psilocybin administration;
4. Have hypertension using the standard criteria of the American Heart Association (values of 140/90 or higher assessed on three separate occasions;
5. History of seizure disorder;
6. Uncontrolled insulin-dependent diabetes;
7. Recent stroke, intracranial or subarachnoid hemorrhage (< 1 year from signing of informed consent form [ICF]), recent myocardial infarction (< 1 year from signing of ICF), clinically significant arrhythmia (< 1 year from signing of ICF);
8. Have liver disease with the exception of asymptomatic subjects with Hepatitis C who have previously undergone evaluation and successful treatment;
9. Lifetime history of substance-induced psychosis;
10. Lifetime history of substance use disorder with a hallucinogen;
11. History of alcohol use disorder in the past 3 months.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility and tolerability | Up to 16 weeks
  Recruitment rate, withdrawal rate, adherence rate, data completion rate, percentage of participants with severe adverse events.

SECONDARY OUTCOMES:
Clinician-Administered PTSD Scale for DSM-5 (CAPS-5) total score | Up to 16 weeks
  The CAPS-5 is a semi-structured clinical interview used to assess index history of DSM-5-defined traumatic event exposure, including the most distressing event, time since exposure, and total number of exposures, as well as frequency and severity of posttraumatic stress symptoms.
Posttraumatic stress disorder Checklist-5 (PCL-5) | Up to 16 weeks
  The PCL-5 is self-report questionnaire in which respondents indicate the presence and severity of PTSD symptoms, derived from the DSM-5 symptoms of PTSD.
Patient Health Questionnaire-9 (PHQ-9) | Up to 16 weeks
  The PHQ-9 is a self-rated measure of depressive symptom severity in the past two weeks. Each of the nine items is rated on a Likert scale, ranging from 0 (not at all) to 3 (nearly every day), and summed for a total score between 0 (no symptoms) to 27 (most severe).
Generalized Anxiety Disorder Scale, 7-item (GAD-7) | Up to 16 weeks
  Total score ranges from 0 to 21; a higher score denotes greater symptom severity.
Dissociative Experiences Scale II (DES-II) | Up to 13 weeks
  The Dissociative Experiences Scale II is a 28-item, self-report measure of dissociative experiences.
Pittsburgh Sleep Quality Index (PSQI) | Up to 13 weeks
  The PSQI is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval.
World Health Organization Well-Being Index, 5-item (WHO-5) | Up to 16 weeks
  The WHO-5 is a measure of overall well-being, rated on a scale of 0 to 25, with higher scores denoting higher quality of life.
Quality of relationships inventory (QRI) | Up to 13 weeks
  The QRI is a self-report questionnaire used to determine the quality relationships consisting of 25 items that are evaluated on a 4-point Likert scale ranging from 1 = not true to 4 = almost always true.
Inventory of psychosocial functioning (IPF) | Up to 13 weeks
  The IPF is an 80-item self-report instrument measuring PTSD-related functional impairment in the past 30 days.
Posttraumatic Maladaptive Beliefs Scale (PMBS) | Up to 13 weeks
  The PMBS is a 15-item scale that was developed to measure maladaptive beliefs about life circumstances that may occur following trauma exposure.
Brief Experiential Avoidance Questionnaire (BEAQ) | Up to 13 weeks
  The BEAQ is a 15-item self-report measure of experiential avoidance.
24-items Multidimensional Psychological Flexibility Inventory (MPFI-24) | Up to 13 weeks
  The MPFI-24 is a 24-item self-report scale developed to assess the specific components of psychological flexibility and inflexibility.
Working Alliance Inventory- Short Form (WAI-SF) | Up to Day 7
  The WAI-SF is a patient-rated measure of the alliance between a therapist and client.
Difficulties in Emotion Regulation Scale-Short Form (DERS-SF) | Up to 13 weeks
  The DERS-SF is an 18-item measure used to identify emotional regulation issues in adults.
Self-Compassion Scale-Short Form (SCS-SF) | Up to 13 weeks
  The SCS-SF is a 12-item self-report measure of self-compassion.
Psychological Insight Questionnaire (PIQ) | Up to Day 3
  The PIQ is a 23-item self-report measure of acute experiences of insight (e.g. awareness into emotions, behaviors, beliefs, memories, or relationships) after taking a psychedelic.
Emotional Breakthrough Inventory (EBI) | Up to Day 3
  The EBI is a measure of emotional release/breakthrough experienced during the acute psychedelic state.
Altered States of Consciousness Rating Scale (ASC) | Up to Day 3
  The ASC measures altered states of consciousness.
Acceptance/Avoidance-Promoting Experiences Questionnaire (APEQ) | Up to Day 3
  The APEQ is a psychometric self-report tool for measuring aspects of the acute psychedelic experience that are associated with longer-term changes in psychological flexibility.
Childhood Trauma Questionnaire-short form (CTQ-SF) | Screening

OTHER OUTCOMES:
Effect on digital physiological passive data collected through the use of a wearable device | Up to 16 weeks
  Example: sleep, activity

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Unity Health Toronto, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Meshkat S, J Zeifman R, Stewart K, Janssen-Aguilar R, Lou W, Jetly R, Monson CM, Bhat V. Psilocybin-assisted massed cognitive processing therapy for chronic posttraumatic stress disorder: Protocol for an open-label pilot feasibility trial. PLoS One. 2025 Jan 17;20(1):e0313741. doi: 10.1371/journal.pone.0313741. eCollection 2025. PMID 39823496